CLINICAL TRIAL: NCT03474224
Title: Correlation Between IN-TArget Time for Mean Arterial Pressure and Stroke Volume During Major Urological Surgery and Tissue Perfusion: the INTAT Observational Study
Brief Title: Hemodynamic Optimization During Major Urological Surgery
Acronym: INTAT
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, RUSSO ANDREA, Medical Doctor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 1822
Record Dates: First submitted 2018-02-25; First posted 2018-03-22 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Hemodynamic Instability
Keywords: stroke volume; goal directed therapy; major urological surgery; mean arterial pressure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- FloTrac patients: patients belong to this group will be managed with a stroke volume target hemodynamic protocol
  Interventions: Device: Ev1000 Clinical Platform from Edwards Lifesciences

INTERVENTIONS:
Device: Ev1000 Clinical Platform from Edwards Lifesciences — The EV1000 Hemodynamic monitoring platform will be used to guide fluid administration following a volume-based parameter such the stroke volume.

SUMMARY:
In this prospective observational study investigators aim to seek for any possible correlation between the venous to arterial carbon dioxide difference (pCO2 gap) at the end of surgery and the percentage of time spent above a predefined threshold of stroke volume (SV) andn mean arterial pressure (MAP).

DETAILED DESCRIPTION:
During major urological surgery (i.e. cistectomy) investigators will use a minimally invasive hemodynamic monitoring system (Flotrac - Vigileo, Edwards ) to guide fluid therapy and vasopressors administration. More specifically stroke volume target will be defined as the maximum SV after a series of fluid boluses, with a 10% tolerance. MAP was considered adequate if above 65 mmHg. After the induction of anesthesia, then each hour during surgery until the end of surgical procedure investigators will assess the time of adherence to the hemodynamic protocol (in terms of both SV and MAP) and the correspondent pCO2 gap. Investigators expect to find an inverse proportionality between the two parameters explored.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for major urological surgery
* ASA 1-2-3

Exclusion Criteria:

* pregnancy
* obesity with a BMI > 35
* controindications to central venous catheter positioning
* end-stage renal disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for major urological surgery who met the above mentioned inclusion criteria will be enrolled. All patients will belong the only study group in which a target-based hemodynamic protocol will be applied
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-07-28 (Actual)

PRIMARY OUTCOMES:
Correlation between the time-in target of MAP and the pCO2 gap at the end of surgery | an average of 8 hours
  The primary outcome will explore the hypothesis that patient with higher adherence of MAP levels above 65 mmHg will have a lower pCO2 gap at the end of surgery
Correlation between the time-in target of SV and the pCO2 gap at the end of surgery | an average of 8 hours
  The co-primary outcome will explore the hypothesis that patient with higher adherence of SV within the maximum value with a 10% tolerance, will have a lower pCO2 gap at the end of surgery

SECONDARY OUTCOMES:
incidence of postoperative overall complications | up to 30 days
  investigators will assess the impact of the intraoperative hemodynamic optimization on the rate of postoperative complications
duration of hospitalization | an average of 2 weeks
  investigators will prospectively evaluate the association between an intraoperative goal-directed fluid therapy with the long of stay

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Russo, MD, Principal Investigator — Department of Anesthesiology
Locations (1):
- Andrea Russo, Rome, Italy